CLINICAL TRIAL: NCT06257511
Title: Developing an Intervention to Improve the Non-Technical Skills of the Cardiac Surgical
Brief Title: Developing an Intervention to Improve the Non-Technical Skills of the Cardiac Surgical Teams
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher left university before the start of recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: K99_01
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-01

CONDITIONS: Patient Care Team; Coronary Artery Disease; Coronary Artery Bypass; Surgery; Hemorrhage Postoperative
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Hemorrhage

STUDY DESIGN:
Intervention Model Description: The goal of this project is to develop and test an intervention to improve the non-technical skills of cardiac surgical teams. The Investigators will develop, pilot test, refine, and assess the preliminary effectiveness of Non-Technical Skills for cardiac Surgery (NOTSCS) intervention on the non-technical skills of participants, operating room (OR) time, and patient post-operative complications (intraoperative bleeding, and unplanned return to the OR.
  Investigators will compare the outcomes between the intervention and control groups, before and after the intervention.
Who Masked: Outcomes Assessor
Masking Description: Investigators will record videos of the participants during simulation sessions, before and after the interventions. The people assessing the non-technical skills of the cardiac surgical teams will be masked if the videos were recorded before or after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Technical Skills for Cardiac Surgery (NOTSCS) intervention group (Experimental): These are the members of the cardiac surgical teams who will be trained in the non-technical skills.
  Interventions: Behavioral: Simulation-Based Mastery Learning of the Non-technical skills
- Control group (No Intervention): These are members of the cardiac surgical teams who will not participate in the intervention.

INTERVENTIONS:
Behavioral: Simulation-Based Mastery Learning of the Non-technical skills — Participants will participate in a simulation-based mastery learning of the non-technical skills.
  Arms: Non Technical Skills for Cardiac Surgery (NOTSCS) intervention group

SUMMARY:
Teams of several medical professionals conduct high-risk cardiac surgical procedures. These professionals work in complex, stressful operating room environments requiring effective communication and teamwork skills. Surgeons, anesthesiologists, perfusionists, nurses, and surgical technicians working in this environment are also vulnerable to human errors. Non-technical skills for surgeons (NOTSS), defined as cognitive skills (situation awareness, decision making) and social skills (leadership, communication, and teamwork) underpinning medical knowledge and technical skills, are essential contributors to better cardiac surgery outcomes. Yet most of the surgical education programs focus only on technical skills, and interventions to improve the non-technical skills of cardiac surgical teams are scarce. The proposed research will develop and pilot-test and evaluate the preliminary effectiveness of an intervention to improve the non-technical skills of cardiac surgical teams.

DETAILED DESCRIPTION:
Over 290,000 Coronary Artery Bypass Graft (CABG) and valve replacement surgeries are performed in the US annually. Around 30% of patients undergoing CABG experience a complication. Notably, hospitals and surgeons with high CABG and valve surgery volumes are more likely to achieve better outcomes. In other surgical specialties, more than 50% of surgical complications are attributable to ineffective non-technical skills for surgeons (NOTSS), defined as cognitive skills (situation awareness, decision making) and social skills (leadership, communication, and teamwork) underpinning medical knowledge and technical skills. The previous work and others found that better non-technical skills were associated with improved risk-adjusted rates of any post-operative complication, mortality, return to the operating room, and intraoperative performance. The investigator have also reported that non-technical skills training programs for general surgeons can effectively improve NOTSS and are associated with improved Operating Room (OR) performance metrics, fewer unplanned reoperations, decreased length of hospital stay, and lower mortality rate. Given our prior work, it is likely that Non-Technical Skills for Cardiac Surgery (NOTSCS) are also important contributors to better cardiac surgery outcomes.

Cardiac surgery procedures are technically challenging for the surgeons and physiologically disruptive for patients, e.g. circulatory arrest, cardiopulmonary bypass, with very little physiologic reserve as a result of their cardiac disease. Cardiac surgeries are conducted by different teams each composed for specialized medical professionals working in concert and relieving each other to support creation of new anatomical structures in the heart (surgery team), cardiopulmonary function (anesthesia team), perfusion to vital organs (perfusionist team), transfusion (blood management team), provision of medicines (operating room pharmacy team) and provision of tools and implants (nursing team). The dramatic and unexpected physiologic changes that occur, large number of medical professionals, extreme sub-specialization of medical professionals, ad-hoc nature of the teams, steep hierarchy between medical professionals and participation of learners all make cardiac surgery operating rooms highly stressful environments. Individuals working in this stressful environment are highly vulnerable to human errors that lead to complications. Yet most of the surgical education programs focus only on technical skills, and interventions to improve the non-technical skills of cardiac surgical teams are scarce. Therefore, there is an urgent need to develop tailored, cardiac surgery-specific interventions to improve the NOTSCS and to assess their effect on patient outcomes.

The goal of this K99/R00 is to develop and test an intervention to improve the non-technical skills of cardiac surgical teams. The investigators will develop, pilot test, refine, and assess the effect of a NOTSCS intervention by applying principles of simulation-based mastery learning (SBML). SBML allows learners to deliberately practice skills until they achieve a mastery level. Most importantly, this application will allow for my development as an independent investigator focused on improving NOTSCS, with a long-term goal of improving cardiac surgery outcomes. The aims of this application are:

K99 Aim 1: To adapt existing non-technical skills performance metrics to cardiac surgical teams. The investigators will identify the behavioral markers required to enhance intraoperative non-technical skills performance for the cardiac surgery teams at academic and community hospitals.

K99 Aim 2: To adapt refine and pilot test an existing NOTSS improvement intervention for cardiac surgery-specific skills, environments, and teams, and assess barriers and facilitators to its implementation.

R00 Aim 1: To assess the preliminary effectiveness of NOTSCS on OR times and patient outcomes.

The research team will implement the NOTSCS intervention to cardiac surgical teams from two academic hospitals. The hypothesis is that a non-technical skills improvement program will be associated with increased NOTSS behaviors, decreased OR time, cardiopulmonary bypass time, time on/off pump, intraoperative bleeding requiring transfusion, and unplanned return to the operating room.

R00 Aim 2: To examine implementation acceptability, feasibility, appropriateness of a SBML NOTSCS intervention. Using quantitative and qualitative feedback, the investigators will map barriers and facilitators to an implementation framework to address barriers to the NOTSCS intervention.

ELIGIBILITY:
Inclusion Criteria:

* All members of the cardiac surgical teams will be eligible to participate in the study (cardiac surgeons, OR nurses, perfusionists, anesthetists...

Exclusion Criteria:

* Clinicians who are not directly involved in intraoperative care of cardiac surgical patients ( for example nurses working only in the recovery room, ICU, floor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Non-technical skills behaviors of the members of the cardiac surgical teams | Non-technical skills will be measured before the intervention, immediately after the intervention, and six months after the intervention
  Investigators will use the Non-Technical Skills for Surgery (NOTSS) rating tool to evaluate the effectiveness of the non-technical skills educational intervention on participants' intraoperative non-technical skills.

SECONDARY OUTCOMES:
Intraoperative performance of the cardiac surgical teams | For each of the cardiac surgeons who will participate in the study, the investigators will compare baseline data (six months collected before implementing the NOTSCS intervention), with data collected after the NOTSCS intervention (six months data).
  Investigators will measure the length of the operation, the length cardiopulmonary bypass time, time on/off pump.
Rate of patients with patients with intraoperative bleeding requiring transfusion, and unplanned return to the operating room | Data for six months before and six months after the intervention
  intraoperative bleeding requiring transfusion, and unplanned return to the operating room. Investigators will conduct a quasi-experimental study. Investigators will compare baseline data (six months collected before implementing the NOTSCS intervention), with data collected after the NOTSCS intervention (six months data).

IPD SHARING:
Plan to Share IPD: Yes
The findings from this study will be at national and international conferences. Additionally, the study team will publish findings from this study in the peer-reviewed scientific journals. Along with publication, cardiac surgery-specific non-technical skills assessment tools, simulation scenarios, and debriefing templates that will be developed in this study, will be shared with the scientific community so that they can understand the process of developing and implementing this project, and possibly replicate it if they are interested. The datasets and coding book, and STATA codes will be shared to the scientific community.
  Quantitative data generated from this project will be made available as soon as the article gets published online. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon completion of the study
Access Criteria: Data will be shared upon contacting the PI